CLINICAL TRIAL: NCT02171377
Title: Quadricipital Electrical Stimulation in COPD Patients Rehabilitation
Acronym: Reha-Res
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/091/HP; 2009-A00665-52 (Registry Identifier: AFSSAPS)
Record Dates: First submitted 2010-10-11; First posted 2014-06-24 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; electrical stimulation; Rehabilitation; exercise test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 : quadricipital electrical stimulation (Experimental): stimulation in addition to rehabilitation (30 min bilateral quadricipital electrical stimulation pd, 5 days per week, 8 weeks)
  Interventions: Device: group 2 : quadricipital electrical stimulation; Device: muscular electrical stimulation
- Group 1 : Pulmonary rehabilitation (Active Comparator): Pulmonary rehabilitation 3 to 5 times per week, 8 weeks
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Device: group 2 : quadricipital electrical stimulation — bilateral quadricipital electrical stimulation 5 sessions a week, (6 - 8 weeks)
  Arms: Group 2 : quadricipital electrical stimulation
Other: pulmonary rehabilitation — exercise training, 3 to 5 times per week, 8 weeks
  Arms: Group 1 : Pulmonary rehabilitation
Device: muscular electrical stimulation — Bilateral quadricipital electrical stimulation 30 min, 5 times per week, 8 weeks,in addition to pulmonary rehabilitation
  Other Names: Mi-Theta-Pro device (Compex medical SA ; CH - 1024 Ecublens); reference 498000 ; serial number WB100000.
  Arms: Group 2 : quadricipital electrical stimulation
Other: pulmonary rehabilitation — exercise training, 45 min, 3 to 5 times per week, 8 weeks
  Other Names: exercise training
  Arms: Group 1 : Pulmonary rehabilitation

SUMMARY:
Quadricipital electrical stimulation added to respiratory rehabilitation in COPD patients.

Quadricipital electrical stimulation (ES) in chronic obstructive pulmonary disease (COPD) patients has been demonstrated to improve both dyspnea and physical status. The aim of our study is to demonstrate that ES added to respiratory rehabilitation program induces a greater improvement on exercise tolerance in such patients.

Design : 160 patients with severe COPD will be randomly assigned to 2 groups : either rehabilitation program (group 1), either ES and rehabilitation program (group 2). In both groups, rehabilitation program comprises endurance training, 18 - 24 sessions (6 - 8 weeks), health education, global muscular strengthening. In group 2, bilateral quadricipital electrical stimulation 30 min sessions is added 5 days / week.

Subjects : COPD patients with FEV1 < 60% pred, FEV1/VC < 70%, and TLC > 80%, with dyspnea, in stable conditions, and 18 > BMI < 35 kg/m² .

Intervention : 6 min walking distance, incremental exercise test data (aerobic capacity, work rate, ventilatory threshold), physical activity with activity monitor, health related quality of life will be determined before and after training.

Abbreviations : FEV1 = forced expiratory volume in 1 sec; VC = vital capacity; TLC = total lung capacity; BMI = body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Subjects : COPD patients with FEV1 < 60% pred, FEV1/VC < 70%, and TLC > 80%, with dyspnea, in stable conditions, and 18 > BMI < 35 kg/m²

Exclusion Criteria:

* BMI 18 < or > 35 kg/m²
* Pregnant women
* peripheral neuropathy
* cardio respiratory incremental test contra-indication
* evolutive cancer
* cardiac or cerebral pace maker, implanted cardio defibrillator
* no informed consent given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
6 minute walking distance | From 6 to 8 weeks

SECONDARY OUTCOMES:
incremental cardio pulmonary exercise test | From 6 to 8 weeks
  Aerobic capacity, maximal achieved work rate, ventilatory threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Bonnevie T, Gravier FE, Debeaumont D, Viacroze C, Muir JF, Cuvelier A, Netchitailo M, Roy AL, Quieffin J, Marques MH, Medrinal C, Dupuis J, Tardif C. Home-based Neuromuscular Electrical Stimulation as an Add-on to Pulmonary Rehabilitation Does Not Provide Further Benefits in Patients With Chronic Obstructive Pulmonary Disease: A Multicenter Randomized Trial. Arch Phys Med Rehabil. 2018 Aug;99(8):1462-1470. doi: 10.1016/j.apmr.2018.01.024. Epub 2018 Feb 16. PMID 29457998